CLINICAL TRIAL: NCT01733602
Title: Does Transcranial Direct Current Stimulation (tDCS) Enhance Outcomes From Computerised Cognitive Remediation in Patients With Schizophrenia?
Brief Title: tDCS to Enhance Cognitive Training in Schizophrenia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The University of New South Wales (Other)
Responsible Party: Principal Investigator, Melissa Pigot, Research Assistant, The University of New South Wales
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11/188
Record Dates: First submitted 2012-11-26; First posted 2012-11-27 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- active tDCS and cognitive training (Experimental): Transcranial direct current stimulation combined with cognitive training
  Interventions: Device: transcranial direct current stimulation
- sham tDCD and cognitive training (Active Comparator): Sham transcranial direct current stimulation combined with cognitive training
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation

SUMMARY:
The primary aim for the study is to determine whether transcranial direct current stimulation (tDCS) enhances training gains on cognitive training (CT) tasks. Secondary aims are to determine whether tDCS combined with CT causes larger transferable improvements on non-trained tasks (i.e., generalisation effects) and whether these generalisation effects are maintained over time (i.e., maintenance effects).

Specific hypotheses are:

1. CT combined with active tDCS will produce greater training gains on CT tasks compared to a similar control group receiving CT with sham tDCS.
2. CT combined with active tDCS will produce greater generalisation effects on non-trained cognitive tasks compared to CT with sham tDCS.
3. The cognitive improvements gained by patients from both interventions will be maintained over 1 month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are 18 years of age or above.
2. Subjects meet criteria for a DSM -IV schizophrenia or schizoaffective disorder but with a stable mental status as demonstrated by a stable Positive and Negative Symptom Score (PANSS) score over a period of 2 weeks.
3. Subjects have had no medication changes in the 2 weeks prior to obtaining informed consent.
4. Subjects are right-handed.
5. Subjects able to give informed consent for the trial.

Exclusion Criteria:

1. Drug or alcohol abuse or dependence (preceding 3 months).
2. Concurrent anticonvulsant or long acting benzodiazepine medication, as these medications may interfere with the effects of tDCS.
3. Subject requires a rapid clinical response due to inanition, psychosis or high suicide risk.
4. Clinically defined neurological disorder or insult, including history of seizures, cerebral aneurysm or trauma, significant head trauma with loss of consciousness for ≥ 30 minutes.
5. Subject has metal in the cranium, skull defects, or skin lesions on scalp at proposed electrode sites.
6. Female subject of child bearing age, sexually active and not using reliable contraception

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2012-11; Primary Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Progression score on cognitive training task. | Post treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Mental Health Rehabilitation Unit (MHRU) at the Sutherland hospital, Sydney, New South Wales, Australia